CLINICAL TRIAL: NCT02277353
Title: Evaluation of Stroke Volume Variation Derived From NICOM as a Predictor of Fluid Responsiveness in Prone Position During Spine Surgery
Brief Title: Evaluation of SVV From NICOM as a Predictor of Fluid Responsiveness in Prone Position During Spine Surgery
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hwan Lee, Assistant Professor, Samsung Medical Center
Other Study IDs: 2014-05-090-003
Record Dates: First submitted 2014-10-09; First posted 2014-10-29 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Fluid Responsiveness; Prone Position; Non Invasive Cardiac Output Monitoring
Keywords: Fluid responsiveness; NICOM; Prone Position; Stroke Volume Variation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All enrolled patients: This study enrolls patients undergoing elective spine surgery in prone position and all enrolled subjects may receive fluid loading with hemodynamic monitoring by Flotrac/Vigileo and NICOM, but the investigator does not assign specific interventions to the subjects of the study because this is a prospective observational study.
  Interventions: Other: Fluid loading to evaluate fluid responsiveness

INTERVENTIONS:
Other: Fluid loading to evaluate fluid responsiveness — loading of hydroxyethyl starch 6ml/kg over 10-15min to all patients

SUMMARY:
NICOM® is a recently developed noninvasive cardiac output monitoring device, and indices derived from NICOM® such as SVV has been reported to predict fluid responsiveness in the previous studies. However, its usefulness in prone positioning has not been investigated. Thus, the aim of this prospective observational study is to evaluate the usefulness of stroke volume variation (SVV) derived from NICOM® to predict fluid responsiveness in prone patients undergoing spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II patients undergoing spine surgery in prone position

Exclusion Criteria:

* Pre-existing arrhythmic disorders/moderate to severe valvular heart disease/obstructive pulmonary disease (COPD grade >2), left ventricular dysfunction with LV EF less than 50, preoperative need for inotropics or vasopressors
* BMI >30kg/m^2 or <15kg/m^2
* Preoperative serum Cr > 1.3mg/dL
* Patients with coagulopathy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing spine surgery under general anesthesia in prone position
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Stroke volume variation from NICOM® | 5 min after infusion of bolus fluid
  predictability of stroke volume variation from NICOM® for fluid responsiveness

SECONDARY OUTCOMES:
pulse pressure variation and stroke volume variation from Flotrac/Vigileo system | 5 min after infusion of bolus fluid
  Correlation with pulse pressure variation, stroke volume variation from Flotrac/Vigileo system

OTHER OUTCOMES:
TPR (total peripheral resistance), TPRI (total peripheral resistance index) | 5 min after infusion of bolus fluid

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Jin Min, MD, Study Director — Samsung Medical Center
Locations (1):
- Samsung Seoul Hospital, Samsung Medical Center, Seoul, South Korea